CLINICAL TRIAL: NCT04675320
Title: Immuno Monitoring in Patient With Epithelial Ovarian Cancer Eligible to PARP Inhibitors
Acronym: IMMUNOPARP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00036-33
Record Dates: First submitted 2020-12-07; First posted 2020-12-19 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer
Keywords: PARP Inhibitors; immunomonitoring
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 specific blood samples :
  * On the first day of anti-PARP treatment (before taking the first dose)
  * Second month of anti-PARP treatment
  * Fourth month of anti-PARP treatment
  * Sixth month of anti-PARP treatment
  * At relapse or cessation of anti-PARP treatment
  For each blood sample
  * 1 heparinized tube (5 mL) for plasmatheque
  * 1 heparinized tube (5 mL) for immunophenotyping,
  * 4 EDTA tubes (4 x 10 mL) for PBMC collection (cryopreservation).
  * 1 EDTA tube (10mL) for quantification of circulating tumor DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-line epithelial ovarian cancer (30 patients): Maintenance treatment of adult patients with newly diagnosed advanced epithelial ovarian, fallopian tube or primary peritoneal cancer (FIGO stages III and IV) with or without BRCA1/2 mutation who have had a partial or complete response to first-line platinum-based chemotherapy.
  Interventions: Biological: blood samples
- Recurrent epithelial ovarian cancer (20 patients): Single-agent maintenance treatment of adult patients with primary, recurrent, platinum-sensitive epithelial ovarian, fallopian tube or peritoneal cancer who have responded (completely or partially) to platinum-based chemotherapy.
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — Blood sampling during PARP inhibitor therapy

SUMMARY:
This study concerns the creation of a biological collection (blood samples) in patients with Epithelial Ovarian Cancer in in order to describe the immune response with PARP inhibitors.

DETAILED DESCRIPTION:
The aim is to assess the impact of anti-PARP on peripheral immune populations and the amount of DNA circulating; to correlate these data with tumor infiltration, with the initial clinical characteristics and with the clinical course; compare the immunogenic effect of different anti-PARPs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years
2. Patient treated for epithelial ovarian cancer
3. Eligible for anti-PARP therapy and in one of the 2 cohorts below:

   * Cohort 1: Maintenance treatment of adult patients with newly diagnosed advanced epithelial ovarian, fallopian tube or primary peritoneal cancer (FIGO stages III and IV) with or without BRCA1/2 mutation, who have had a partial or complete response to first-line platinum-based chemotherapy.
   * 2nd cohort: single-agent maintenance treatment of adult patients with platinum-sensitive, recurrent primary epithelial ovarian, fallopian tube or peritoneal cancer who have responded (completely or partially) to platinum-based chemotherapy.
4. Patient having signed the informed consent form.
5. Patient fit and able to comply with the protocol for the duration of the study, including visits, scheduled sampling and follow-up.
6. Patient affiliated to the social security system.

Exclusion Criteria:

1. Non-epithelial tumour of the ovary
2. Patient unable to understand, read and/or sign informed consent.
3. Current or previous use of immunosuppressive medication within 14 days prior to inclusion (except intranasal corticosteroids, systemic corticosteroids in physiological doses not exceeding 10 mg daily of prednisone or its equivalent, corticosteroids used as premedication for hypersensitivity reactions.
4. Patient participating in other research that may modify the systemic treatment administered in the cohort in which she will be included.
5. Pregnant or breast-feeding women.
6. HIV and/or HBV and/or HCV serology positive.
7. Patient refusal.
8. Person benefiting from a system of protection for adults (including guardianship, curatorship and safeguard of justice).
9. Inability to undergo medical follow-up for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Cohort 1: Maintenance treatment of adult patients with newly diagnosed BRCA1/2-mutated advanced epithelial ovarian, fallopian tube or primary peritoneal cancer (FIGO stages III and IV) who have had a partial or complete response to first-line platinum-based chemotherapy. BRCA-mutated epithelial ovarian cancer - maintenance with Olaparib / Niraparib or Olaparib + bevacizumab
  * Cohort 2: Single-agent maintenance treatment of adult patients with platinum-sensitive, recurrent primary epithelial ovarian, fallopian tube or peritoneal cancer who are responding (complete or partial) to platinum-based chemotherapy. Recurrent epithelial ovarian cancer - maintenance with Niraparib or Olaparib
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Immune response in plasma | From date of inclusion until the date of first documented progression or date of death from any cause assessed up to 24 months
  Realization of a plasma library
Immune response in PBMC | From date of inclusion until the date of first documented progression or date of death from any cause assessed up to 24 months
  Realization of a PBMC bank
Immune response in tumor DNA | From date of inclusion until the date of first documented progression or date of death from any cause assessed up to 24 months
  Realization of a circulating tumor DNA bank

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU Jean Minjoz, Besançon
  - Centre Georges Francois Leclerc, Dijon